CLINICAL TRIAL: NCT03211676
Title: Comparison of Hemodialysis With Medium Cut-off Dialyzer (Theranova) and High Flux Dialyzer on Removal of Small and Middle Size Molecules, Inflammatory Parameters and Oxidative Stress. An Open Cross Over Randomized Study
Brief Title: Comparison of Hemodialysis With Medium Cut-off Dialyzer (Theranova) and High Flux Dialyzer
Acronym: THERANOVA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2016-A01679-42
Record Dates: First submitted 2017-05-18; First posted 2017-07-07 (Actual); Last update posted 2020-04-13 (Actual); Status verified 2020-04

CONDITIONS: End Stage Renal Disease; Dialysis Related Complication; Dialysis Amyloidosis
Keywords: dialyzer; beta2-microglobilin; myoglobin
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Theranova-500 (Active Comparator)
  Interventions: Device: Theranova-500 dialyzer; Device: Elisio-21H
- Elisio-21H (Sham Comparator)
  Interventions: Device: Theranova-500 dialyzer; Device: Elisio-21H

INTERVENTIONS:
Device: Theranova-500 dialyzer — hemodialysis with Theranova-500 dialyzer.
Device: Elisio-21H — hemodialysis with Elisio-21H dialyzer

SUMMARY:
The aim of this study is to evaluate the removal of midle molecules and inflammatory cytokines with the Theranova-500 ™ dialyzer (medium cut-off membrane, Baxter®) versus a high flux dialyzer Elisio-21H ™ (High-flux membrane, Nipro®) in chronic hemodialysis.

Evaluation of nutritional parameters, inflamatory parameters and oxidative stress will also be carried out.

Finally, the investigators will compare hepcidin levels and the erythropoietin resistance index between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patient suffering from chronic terminal renal failure excluding nephropathy with myelomatous cylinders, hemodialysis for more than 6 months,
* Patient under dialyser Elisio-21H ™ for more than 3 months
* Patient including the protocol scheme and able to comply with it
* Free subject, without guardianship or curatorship or subordination
* Patients benefiting from a Social Security scheme or benefiting from it through a third party
* Non-opposition given by the patient after clear and fair information on the study

Exclusion Criteria:

* Age <18 years
* Patient with an associated pathology (evolutionary cancer, progressive infectious disease or chronic inflammatory disease) that may excessively influence CRP levels (CRP> 60 mg / L)
* Patient following another protocol of research or period of exclusion of another protocol
* Patients not benefiting from a Social Security scheme or not benefiting from it through a third party
* Persons benefiting from enhanced protection, namely minors, persons deprived of their liberty by a judicial or administrative decision, persons staying in a health or social institution, adults under legal protection, and finally patients in emergencies .
* Pregnant or nursing women, women of childbearing age who do not have effective contraception (hormonal / mechanical: oral, injectable, transcutaneous, implantable, intrauterine device, or surgical: tubal ligation, hysterectomy, total ovariectomy ).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2017-06-07 (Actual); Primary Completion 2018-03-14 (Actual); Study Completion 2018-06-14 (Actual)

PRIMARY OUTCOMES:
Removal of myoglobin | After 3 months
  myoglobin Reduction ratio.

SECONDARY OUTCOMES:
Removal of beta2 microglobulin | After 3 months
  Reduction rate and clearances of beta2 microglobulin
Removal of urea | After 3 months
  Reduction ratio and clearances of urea
Removal of creatinine | After 3 months
  Reduction ratio and clearances of creatinine
Removal of interleukin 6 | After 3 months
  Reduction ratio and clearances of interleukin 6
Removal of IL-1beta | After 3 months
  Reduction ratio and clearances of IL-1beta
Removal of TNF alpha | After 3 months
  Reduction ratio and clearances of TNF alpha
Removal of leptin | After 3 months
  Reduction ratio and clearances of leptin
Removal of alpha 1 microglobulin | After 3 months
  Reduction ratio and clearances of alpha 1 microglobulin
Removal of retinol binding protein | After 3 months
  Reduction ratio and clearances of retinol binding protein
Removal of hyaluronic acid | After 3 months
  Reduction ratio and clearances of hyaluronic acid
Removal of FGF 23 (fibroblast growth factor 23) | After 3 months
  Reduction ratio and clearances of FGF 23
Removal of prolactin | After 3 months
  Reduction ratio and clearances of prolactin
Removal of free light chain kappa | After 3 months
  Reduction ratio and clearances of free light chain kappa
Removal of free light chain lambda | After 3 months
  Reduction ratio and clearances of free light chain lambda
comparison of pre dialysis level of hepcidin | After 3 months
  comparison of average of pre dialysis level of hepcidin
comparison of pre dialysis level of superoxide dismutase | After 3 months
  comparison of average of pre dialysis level of superoxide dismutase
comparison of pre dialysis level of isoprostan | After 3 months
  comparison of average of pre dialysis level of isoprostan
comparison of pre dialysis level of human oxidized LDL | After 3 months
  comparison of average of pre dialysis level of human oxidized LDL
comparison of pre dialysis level of albumin | After 3 months
  comparison of average of pre dialysis level of albumin
comparison of pre dialysis level of prealbumin | After 3 months
  comparison of average of pre dialysis level of prealbumin
comparison of post dialysis level of albumin | After 3 months
  comparison of average of post dialysis level of albumin
comparison of level of middle molecules and albumin in the dialysate | After 3 months
  comparison of average level of midlle molecules and albumin in dialysate
comparison of use of erythrpoietin | After 3 months
  Comparison of the erythropoietin resistance index
comparison of hemoglobin levels | After 3 months
  comparison of average of predialysis hemoglobin levels
comparison of pre dialysis level of CRP | After 3 months
  comparison of average of pre dialysis level of CRP
comparison of pre dialysis level of SAA | After 3 months
  comparison of average of pre dialysis level of SAA

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed BELMOUAZ, Principal Investigator — Poitiers University Hospital
Locations (1):
- CHU DE Poitiers, Poitiers, France

IPD SHARING:
Plan to Share IPD: No